CLINICAL TRIAL: NCT00230984
Title: Effects of Home Pulmonary Rehabilitation in Patients With Chronic Respiratory Failure and Nutritional Depletion.
Brief Title: IRAD2 : Patients With Respiratory Failure at Home
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Societe Francophone de Nutrition Enterale et Parenterale (Other); Association ANTADIR , (Unknown); Ministry of Health, France (Other Government); Association AGIR à Dom, (Unknown); Nutricia France, swizerland), (Unknown); Organon (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DCIC 01 05
Record Dates: First submitted 2005-09-30; First posted 2005-10-03 (Estimated); Last update posted 2009-07-08 (Estimated); Status verified 2006-07

CONDITIONS: Chronic Respiratory Failure; Nutritional Depletion
Keywords: Chronic Respiratory Failure; Pulmonary Rehabilitation; Nutritional Depletion; Home; COPD; Oral Dietary Supplements; Therapeutic Education; Androgens; Exacerbation; Survival
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Educational Status; Dietary Supplements; testosterone undecanoate; Menogaril

INTERVENTIONS:
Behavioral: education
Drug: Oral dietary supplements (563 kcal/d), RESPIFOR
Behavioral: exercises on an ergometric bicycle 3 to 5 times a week
Drug: 160 mg/d of oral testosterone undecanoate in men, 80 mg/d in women

SUMMARY:
Title : Effects of home pulmonary rehabilitation in patients with chronic respiratory failure and nutritional depletion.

This is a randomized controlled, open clinical trial with two groups.

* first group, 100 patients : control group, patients followed with no add-on intervention
* Second group, 100 patients : rehabilitation group with education, oral supplements, exercise and androgenic steroids.

DETAILED DESCRIPTION:
Title : Effects of home pulmonary rehabilitation in patients with chronic respiratory failure and nutritional depletion

State of the art :

The IRAD2 trial is evaluating a 3-month home intervention which includes education, oral supplements, exercise and androgenic steroids in undernourished patients with chronic respiratory failure. The main objective is to increase the six-minute walking distance by more than 50 m with an improvement in health-related quality-of-life. Secondary end-points include a reduction in exacerbation rates by 25%, a reduction in health-related costs and an increase in survival during the year following intervention.

Material and methods :

This interventional, multi-centre, prospective, two-armed parallel, controlled trial is being conducted in 200 patients. In both groups, "Control" and "Rehabilitation", 7 home visits are scheduled during the 3-month intervention for education purpose. In the "Rehabilitation" group, patients will receive 160 mg/d of oral testosterone undecanoate in men, 80 mg/d in women, oral dietary supplements (563 kcal/d) and exercises on an ergometric bicycle 3 to 5 times a week.

Expected results :

In the event of significant responses to intervention, this trial would validate a comprehensive and global home-care for undernourished patients with chronic respiratory failure combining therapeutic education, oral supplements, androgenic substitution and physical activity.

ELIGIBILITY:
Inclusion Criteria:

* well informed and consenting person
* woman is old enough to procreate
* Assisted respiratory treatment at home for 3 months : oxygenotherapy > 8 hours per day and/or assisted ventilation > 6 hours per day.
* PaO2 without oxygenotherapy ≤ 8 kPa or 60 mmHg on ambient air at the beginning of assisted respiratory treatment.
* Affection : chronic obstructive bronchopneumopathy, diffuse bronchial dilatation, non neuromuscular restrictive syndrome (pulmonary diffuse infiltration, parietal lesion) obstructive and restrictive syndrome.
* malnourished person, one of following criteria :Body Mass Index ≤ 21kg/m2 or weight loss (10% of the previous weight) or non-fatty mass measured by 50 Hz impedancemetry ≤25th percentiles or ≤ 63% of ideal weight for women, ≤ 67% of ideal weight for men.

Exclusion Criteria:

* Sleep apnea with daytime drowsiness (drowsiness scale of Epworth > 9/24)
* Known pathology that reduce the vital prognosis at 6 months (AIDS, cancer...).
* History of hormone dependent cancer ( breast cancer, prostate cancer), pathologic Prostate Specific Antigen.
* Inability to follow a rehabilitation program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2003-04; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
An increase of the six-minute walking distance by more than 50 m with an improvement in health-related quality-of-life.

SECONDARY OUTCOMES:
Reduction in exacerbation rates by 25%
Quality of life assessed by generic QOL.
Reduction in health-related costs
Increase in survival during the year following intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe PISON, MD, Principal Investigator — Pneumology Department, University Hospital of Grenoble
Locations (8):
- France (7):
  - University Hospital Dominique Larrey, Limoges
  - Rehabilitation Department of Cyr Voisin, Loos
  - University Hospital Arnaud de Villeneuve, Montpellier
  - Hospital la Pitiè-Salpétrière, Paris
  - University Hospital of Poitiers, Poitiers
  - University Hospital Bois Guillaume, Rouen
  - North University Hospital of St Etienne, Saint-Etienne
- Departement of Medicine, University Hospital of Genève, Geneva, Switzerland

REFERENCES:
- [Background] Veale D, Chailleux E, Taytard A, Cardinaud JP. Characteristics and survival of patients prescribed long-term oxygen therapy outside prescription guidelines. Eur Respir J. 1998 Oct;12(4):780-4. doi: 10.1183/09031936.98.12040780. PMID 9817145
- [Background] Ronning O. Alterations in craniofacial morphogenesis induced by parenterally administered papain. An experimental study on the rat. Suom Hammaslaak Toim. 1971;67:Suppl 3:3-96. No abstract available. PMID 5292850
- [Background] Chailleux E, Fauroux B, Binet F, Dautzenberg B, Polu JM. Predictors of survival in patients receiving domiciliary oxygen therapy or mechanical ventilation. A 10-year analysis of ANTADIR Observatory. Chest. 1996 Mar;109(3):741-9. doi: 10.1378/chest.109.3.741. PMID 8617085
- [Background] Long term domiciliary oxygen therapy in chronic hypoxic cor pulmonale complicating chronic bronchitis and emphysema. Report of the Medical Research Council Working Party. Lancet. 1981 Mar 28;1(8222):681-6. PMID 6110912
- [Background] Okubadejo AA, Paul EA, Jones PW, Wedzicha JA. Does long-term oxygen therapy affect quality of life in patients with chronic obstructive pulmonary disease and severe hypoxaemia? Eur Respir J. 1996 Nov;9(11):2335-9. doi: 10.1183/09031936.96.09112335. PMID 8947081
- [Background] Barnes PJ. Novel approaches and targets for treatment of chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 1999 Nov;160(5 Pt 2):S72-9. doi: 10.1164/ajrccm.160.supplement_1.17. PMID 10556174
- [Background] Hunter AM, Carey MA, Larsh HW. The nutritional status of patients with chronic obstructive pulmonary disease. Am Rev Respir Dis. 1981 Oct;124(4):376-81. doi: 10.1164/arrd.1981.124.4.376. PMID 6794394
- [Background] Schols AM, Soeters PB, Dingemans AM, Mostert R, Frantzen PJ, Wouters EF. Prevalence and characteristics of nutritional depletion in patients with stable COPD eligible for pulmonary rehabilitation. Am Rev Respir Dis. 1993 May;147(5):1151-6. doi: 10.1164/ajrccm/147.5.1151. PMID 8484624
- [Background] Schols AM. Nutrition in chronic obstructive pulmonary disease. Curr Opin Pulm Med. 2000 Mar;6(2):110-5. doi: 10.1097/00063198-200003000-00005. PMID 10741769
- [Background] Schols AM, Mostert R, Soeters PB, Greve LH, Wouters EF. Nutritional state and exercise performance in patients with chronic obstructive lung disease. Thorax. 1989 Nov;44(11):937-41. doi: 10.1136/thx.44.11.937. PMID 2595635
- [Derived] Pison CM, Cano NJ, Cherion C, Caron F, Court-Fortune I, Antonini MT, Gonzalez-Bermejo J, Meziane L, Molano LC, Janssens JP, Costes F, Wuyam B, Similowski T, Melloni B, Hayot M, Augustin J, Tardif C, Lejeune H, Roth H, Pichard C; IRAD Investigators. Multimodal nutritional rehabilitation improves clinical outcomes of malnourished patients with chronic respiratory failure: a randomised controlled trial. Thorax. 2011 Nov;66(11):953-60. doi: 10.1136/thx.2010.154922. Epub 2011 Jun 23. PMID 21700760